CLINICAL TRIAL: NCT03450460
Title: A Randomized Controlled Feasibility Trial on the Ontario Brain Injury Association Peer Support Program
Brief Title: Ontario Brain Injury Association (OBIA) Peer Support Program
Acronym: TOPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Rehabilitation Institute (Other)
Collaborators: Ontario Neurotrauma Foundation (Other); Ontario Brain Injury Association (Unknown)
Responsible Party: Principal Investigator, Sarah Munce, Scientist, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TorontoRI
Record Dates: First submitted 2018-02-22; First posted 2018-03-01 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Acquired Brain Injury
Keywords: peer support; feasibility trial; mixed methods
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1/week peer support (Experimental): These individuals with acquired brain injury will receive the Ontario Brain Injury Association Peer Support program once per week.
  Interventions: Behavioral: Peer support
- wait list control group (No Intervention): These individuals with acquired brain injury will receive the Ontario Brain Injury Association Peer Support once the trial period is complete.

INTERVENTIONS:
Behavioral: Peer support — The Program matches volunteer Mentors and Partners for a series of one-to-one interactions that focus on the discussion and resolution of problems or issues (i.e., problem solving) related to one or several key topic areas including family and friends, resources, life changes or challenges, (health care) professionals, social/recreational activities, work/employment/training/volunteering, the brain injury itself, emotions or feelings, and other issues.27 Once the match is established, the Mentor and Partner communicate with one another primarily by telephone until the problems or issues are either resolved or a referral to another service is made (i.e., counselling or community support services). For some partnerships, communication by email or video conferencing is used.27 Most telephone calls last between 20 and 40 minutes (personal communication) and are held weekly.
  Arms: 1/week peer support

SUMMARY:
Most people with moderate or severe TBI have difficulty returning to their usual social roles and activities. The OBIA has developed a program where peers (other individuals living with TBI) coach or mentor those with more recent brain injury. The objective of this project is to evaluate the feasibility of measuring the impact of the OBIA Peer Program on social participation and mood compared to a control group who have not received peer support yet.

The proposed study will involve three phases. It will begin with a qualitative component (stakeholder interviews), then a pilot RCT, and end with more interviews to explore the success of the study intervention. A qualitative descriptive approach will be used at these first and last phases of the study. In Phase 1, interviews will be conducted with approximately 15 participants including individuals with moderate to severe TBI, caregivers, Mentors, OBIA staff members, and health researchers. The proposed Phase 2 will be a clinical trial, conducted with 60 participants. These participants will be randomized to one of three groups: a twice a week Program (n=20), a once a week Program (n=20), or the wait list control group (n=20). For Phase 3, a sub group of approximately 25 participants from Phase 2 who participated in the OBIA Peer Support Program will be asked to participate in a one-on-one, telephone/Skype interview. A sub-group of Mentors will also be asked to participate in a one-on-one, telephone/Skype interview.

This research project will address the highest priority areas of "strategies to enhance social participation and community life (personal relationships)" and "psychological strategies to improve mood, depression, and irritability", as identified in the ONF's Request for Proposals on "Addressing Evidence Gaps in Moderate to Severe TBI Rehabilitation". The study will provide important results to inform a RCT (of appropriate size) on the impact of peer support on the social participation and mood of individuals with moderate to severe TBI. This study will then provide the best evidence to support the recommendation on "a peer-supported relationship model of intervention", and inform future versions of the INESSS-ONF Guideline.

DETAILED DESCRIPTION:
Phase 1 - Understanding the Enablers, Barriers of Implementing the Trial Protocol

Specific Objective: To understand the perceived enablers and barriers of implementing the peer support trial protocol, including the perceived enablers and barriers to participant recruitment, retention, adherence, and data collection, of implementing the selected outcomes measures, and of participating in the trial, from the perspective of stakeholders (knowledge users) including individuals with moderate to severe TBI, caregivers, OBIA Peer Support Program Mentors, OBIA staff members who are a part of the Peer Support Program, health services and knowledge translation (KT) researchers with expertise in TBI, and methodologists with expertise in clinical trials; Hypothesis: A better understanding of the perceived enablers and barriers of implementing the peer support trial protocol will enhance the effectiveness of the intervention and feasibility of the trial in Phase 2 and results will be used to refine the research protocol for the RCT, if necessary.

Participants and recruitment: A purposive sampling of each of the different stakeholder groups will be used. The OBIA Peer Support Program Database will be used to recruit the Partners (including caregivers) and Mentors. On-line searches and/or the contacts of the Principal Investigators will be used to recruit the OBIA staff members and the researchers/methodologists. We will aim to recruit a total of 15 key informants for Phase 1. Individuals who are interested in participating in the study will contact the Research Coordinator via telephone or email to gain further information about the study. The eligibility criteria of all participants will be confirmed by the Research Coordinator. This process will be followed for all phases of the study.

Data collection: participants will take part in a one-on-one, semi-structured telephone/Skype interview lasting approximately 45-60 minutes. All interviews will be digitally recorded and transcribed verbatim for data analysis. During transcription, any identifying information will be removed and the participant will be assigned a coded identifier.

Data analysis: analysis will be conducted using inductive thematic analysis as described by Braun and Clark (2006). The analysis will assess the perceived enablers and barriers to participant recruitment, retention, adherence, and data collection, of implementing the selected outcomes measures, and of participating in the OBIA Peer Support Program and the trial itself. To facilitate the organization and analysis of the qualitative data, the Principal Investigator's/Research Coordinator's reflective notes from the interviews, as well as the transcripts, will be entered into NVivo v.11.

Phase 2 - Evaluating the Feasibility of the Trial Protocol, Conducting a (Pilot) Randomized Controlled Feasibility Trial

Specific Objective: a) To evaluate the feasibility of participant recruitment and retention, data collection, as well as participant adherence to the OBIA Peer Support Program; b) To estimate effect sizes of the immediate impact of the twice/week versus once/week OBIA Peer Support Program compared to a wait list control group on social participation (primary outcome), mood, HRQoL, and self-efficacy (secondary outcomes); Hypotheses: a) It is expected that adequate (i.e., ≥75%) recruitment, retention and adherence to the OBIA Peer Support Program will be achieved; b) It is expected that the six-month OBIA Peer Support Program delivered twice weekly will lead to greater mean improvement, on measures of social participation, mood (i.e., depressive symptoms), HRQoL, and self-efficacy, than the same program delivered once weekly or a wait list control intervention (i.e., a dose response effect will be observed); c) It will be possible to estimate the magnitude of effect to allow the sample size calculation for a definitive trial; Significance: The results of the currently proposed research will support a future definitive RCT.

Participants and recruitment: eligible Partner participants will include community-based (i.e., no longer participating in a comprehensive rehabilitation program) individuals who have a moderate to severe TBI. Partners will be recruited via an online advertisement posted on the OBIA website as well as the websites of the 14 participating brain injury associations. Mentor participants may also be recruited from the OBIA Peer Support Program Database. We will aim to recruit a total of 60 Partners (i.e., n=20 participants per group) and 20-40 Mentors (those paired with partners in the intervention arm) for Phase 2.

Intervention and Control Groups: Participants in the intervention groups will take part in the OBIA Peer Support Group, receiving either twice a week (i.e., two 20-40 minute calls) or once a week (i.e., one 20-40 minute call) support. In keeping with an average duration of support, and for the purposes of the currently proposed study, the intervention duration will be 6 months. Participants in the control group will be assigned to a wait list. They will receive the OBIA Peer Support Program after the intervention group (i.e., after 6 months). This assignment does not represent a significant variation in the usual intake procedure, as the OBIA Peer Support Program already maintains a wait list (personal communication).

Sample Size, Randomization, and Blinding: since this is a feasibility study, a formal sample size calculation will not be performed. The recruitment of 20 participants in each arm of the trial is judged to be feasible and will produce a robust and useful amount of data. Partner participants who meet the inclusion and exclusion criteria and have provided informed consent to take part in the trial will be randomized to either the intervention (twice/week or once/week Program) or the wait list control groups. Mentors will be assigned to those randomized into the intervention arms by the OBIA Peer Support Program using their usual methods. A web-based randomization service with secure password protected login using random variable block-size will be used. Due to the nature of the intervention, blinding of the Partners and Mentors will not be possible. However, the processes of outcome assessment and data analysis will be blinded.

Data collection: baseline data including demographic and descriptive information (e.g., age, sex, severity of injury, marital status), as well as the following outcomes measures described below, will be captured prior to randomization: social participation using the Community Integration Questionnaire (CIQ); mood (i.e., depressive symptoms) using the nine-item Patient Health Questionnaire (PHQ-9); health-related quality of life (HRQoL) using the Short Form-12 Health Survey (SF-12); self-efficacy using the TBI Self-efficacy Questionnaire. Follow-up assessments for the outcome measures will occur at 6 weeks, 3 months, and 6 months. Participants will have the option to complete their baseline demographic and descriptive information and outcome measures as well as their follow-up assessments themselves (i.e., paper-based and mailed back to the research team), by telephone, or on-line via Survey Monkey®.

Data analysis: Quantitative Component: baseline characteristics (e.g., age, sex, severity of injury, marital status, etc.) will be described and any differences between the three groups will be compared using means/medians and frequencies and proportions. As this is a feasibility study, and the ability to collect data is being tested, no data imputation will be performed to account for missing data. The feasibility of recruitment will be based on whether 60 participants (i.e., 20 participants in each arm of the trial) can be enrolled in the trial during the 6-month recruitment period. The number of individuals who provide informed consent per month will also be calculated. The feasibility of retention will be assessed by calculating the proportion of participants with complete data on each outcome measure at 6 weeks, 3 months, and 6 months. To evaluate participant adherence, the proportion of twice-weekly and weekly sessions attended by the participants will be calculated. The proportion of participants who withdraw from the intervention at 6 weeks, 3 months, and 6 months will be calculated along with the reason(s) for withdrawing. The feasibility threshold will be set at >75% for recruitment, retention, and adherence (to the intervention). To evaluate changes between groups, the analysis plan will focus on mean change scores and confidence intervals (i.e., mixed-design analysis of variance model) for the outcome measures described above. Effect sizes will be calculated via Cohen d to reflect the impact of the OBIA Peer Support Program on social participation, mood, HRQoL, and self-efficacy.

UPDATE TO PHASE 2 AFTER COMPLETING PHASE 1

After the completion of the phase 1 study and prior to implementing the phase 2 pilot RCT, the following procedures were changed/finalized for the RCT: 1) the study will only include the once/week intervention arm and a wait-list control (participant recruitment expectations adjusted accordingly to 40 partners (20 per arm) and 20 mentors (to be matched with those in the intervention arm); 2) the trial length has been reduced from 6 months to 4 months, and data collection points now include baseline, 2 months, and 4 months; 3) The Short Form-20 Health Survey (SF-20) will replace the SF-12 outcome measures; and, 4) data collection will be done by telephone.

Phase 3 - Exploring the Impact and Acceptability of the OBIA Peer Support Program and the Trial Protocol

Specific Objective: To explore the impact and acceptability of the OBIA Peer Support Program and the trial itself from the perspective of Partners and Mentors; Hypothesis: It is expected that the OBIA Peer Support Program will be acceptable to both the Partners and Mentors and that an increased understanding of the OBIA Peer Support Program and the trial itself will be achieved; Significance: The results of Phase 3 will lead to an understanding of the "active ingredients" or mechanisms that are associated with improved outcomes and the impact of "dosage" of interactions. Furthermore, the results of Phase 3 will refine and improve future iterations of the OBIA Peer Support Program and the implementation of the definitive RCT.

Participants and recruitment: Purposive sampling will be used to recruit intervention group Partner participants in Phase 3 (e.g. to ensure participants with a range of severity of TBI), and all prticipating Mentors will be approached about participating in the interviews. Recruitment of participants will cease once data saturation has been achieved, which is the point when successive interviews become repetitive and no new responses or themes emerge. We will aim to recruit a total of 25 Partners and Mentors for Phase 3.

Data collection: participants will take part in a one-on-one, semi-structured telephone/Skype interview lasting approximately 45-60 minutes about their experience with the RCT. All interviews will be digitally recorded and transcribed verbatim for data analysis. During transcription, any identifying information will be removed and the participant will be assigned a coded identifier.

Analysis Plan: analysis will be conducted using inductive thematic analysis as described by Braun and Clark (2006) and will assess participants' experiences with the intervention and the trial protocol itself (i.e., the impact and acceptability of the program itself/intervention and the trial protocol itself). To facilitate the organization and analysis of the qualitative data, the Principal Investigator's/Research Coordinator's reflective notes from the interviews, as well as the transcripts, will be entered into NVivo v.11.

ELIGIBILITY:
For Phase 1

Inclusion Criteria

Partner participants, including caregiver Partners,

* Community-based (i.e., no longer participating in a comprehensive rehabilitation program) individuals;
* Have a moderate to severe TBI (Glasgow Coma Scale ≤12) or have cared for (i.e., unpaid) an individual with moderate to severe TBI for at least one year;
* Are 18 years of age or older;
* Have participated in the OBIA Peer Support Program;
* Are fluent in English; and,
* Are able to provide informed consent/have an available proxy who is able to provide informed consent.

Mentor participants -Completed at least one partnership with the OBIA Peer Support Program

Exclusion Criteria

Partner participants, including caregiver Partners,

-Individuals who are medically unstable or have active suicidal ideation

For Phase 2 and 3

Inclusion Criteria

Partner/Mentor participants

* Community-based (i.e., no longer participating in a comprehensive rehabilitation program);
* Have a moderate to severe TBI (Glasgow Coma Scale of 12 or less);
* Are 18 years of age or older;
* Are fluent in English; and,
* Are able to provide informed consent/have an available proxy who is able to provide informed consent.

  * Note that Mentor participants may include newly-trained Mentors or Mentors that have already had previous mentorship experience with the OBIA Peer Support Program.

Exclusion Criteria

* Previously participated in the OBIA Peer Support Program or currently receiving peer support/self-management program elsewhere;
* Are medically unstable; and,
* Have active suicidal ideation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 13 (Actual)
Dates: Start 2018-05-16 (Actual); Primary Completion 2020-02-13 (Actual); Study Completion 2020-06-18 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Participation at 4 months | Baseline to 4 months
  Community Integration Questionnaire (CIQ)

SECONDARY OUTCOMES:
Change from Baseline Mood at 4 months | Baseline to 4 months
  Patient Health Questionnaire-9
Change from Health-related Quality of Life at 4 months | Baseline to 4 months
  Short-Form-20 Health Survey
Change from Self-efficacy at 4 months | Baseline to 4 months
  Traumatic Brain Injury Self-efficacy Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Munce, Principal Investigator — Toronto Rehabilitation, University Health Network
Locations (1):
- Ontario Brain Injury Association, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Munce SEP, Jaglal S, Kastner M, Nelson MLA, Salbach NM, Shepherd J, Sweet SN, Wilcock R, Thoms C, Bayley MT. Ontario Brain Injury Association Peer Support Program: a mixed methods protocol for a pilot randomised controlled trial. BMJ Open. 2019 Mar 23;9(3):e023367. doi: 10.1136/bmjopen-2018-023367. PMID 30904839